CLINICAL TRIAL: NCT06711237
Title: Comparison of Two Different Excess Cement Clean-up Options for Cementing Metal-free Ceramic Restorations on Dental Implants
Brief Title: Resin-Cement Type Influence on Cement Remnants in Implant-Supported Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vilniaus Implantologijos Centro (VIC) Klinika (Network)
Collaborators: Harvard School of Dental Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: VIC1
Record Dates: First submitted 2024-11-24; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Dental Cements
Keywords: cemented restoration; implant-supported fixed dental prosthesis; cement remnants; peri-implant health

STUDY DESIGN:
Intervention Model Description: sequential design with a washout period
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Self-Adhesive Resin Cement (RC) (Experimental): Single-unit implant-supported single crowns were cemented to the abutments using a self-adhesive resin cement (RC). Residual cement was removed, and the restorations were retrieved for analysis of cement remnants.
  Interventions: Other: self-adhesive resin cement (RC); Other: resin-modified glass-ionomer cement (RMGIC)
- Resin-modified Glass-Ionomer Cement (RMGIC) (Experimental): Single-unit implant-supported single crowns were cemented to the abutments using a resin-modified glass-ionomer cement (RMGIC). Residual cement was removed, and the restorations were retrieved for analysis of cement remnants.
  Interventions: Other: self-adhesive resin cement (RC); Other: resin-modified glass-ionomer cement (RMGIC)

INTERVENTIONS:
Other: self-adhesive resin cement (RC) — Single-unit implant-supported single crowns were cemented to the abutments using a self-adhesive resin cement (RC). Residual cement was removed, and the restorations were retrieved for analysis of cement remnants.
Other: resin-modified glass-ionomer cement (RMGIC) — Single-unit implant-supported single crowns were cemented to the abutments using a resin-modified glass-ionomer cement (RMGIC). Residual cement was removed, and the restorations were retrieved for analysis of cement remnants.

SUMMARY:
This study quantitatively compared cement residues of two resin cement types around implant-supported restorations (ISR) with a crown-abutment margin located at the gingival level. This prospective, single-blinded, cross-over clinical trial compared optically detectable cement remnants between Self-Adhesive Resin Cement (RC) and Resin-Modified Glass Ionomer Cement (RMGIC).

DETAILED DESCRIPTION:
This prospective, two-arm, non-randomized, clinical trial compared detectable cement remnants on 30 patients and 60 ISR. Two cements were compared; self-adhesive resin (RC) and resin-modified glass ionomer (RMGIC). Comparisons were carried out on identical pairs of ISR tested within the same patients with a 1-week healing interval. The primary outcome variable was the ratio of cement-covered area to total crown area. Areas were analyzed ex-situ by standardized digital image analysis.

ELIGIBILITY:
Inclusion Criteria:

* physical and psychological ability to undergo implant therapy (ASA I or II)
* presence of a single mandibular molar indicated for extraction with adjacent healthy and present natural teeth or implant-supported restoration
* presence of ≥ 6 mm width and ≥ 10 mm height native bone ridge - presence of intact alveolar bone walls after tooth extraction and presence of interradicular bone > 4 mm to achieve primary implant stability
* presence of ≥ 1.5 mm distance to adjacent teeth at the bone level
* overall healthy, non-inflamed keratinized soft tissues.

Exclusion Criteria:

Presence of general conditions contributory to dental implant treatment comprising but not limited to:

* presence of active periodontitis 25
* poor oral hygiene as determined by the Oral Health Index (OHI)
* pregnant or lactating
* presence of uncontrolled medical systemic conditions, e.g. diabetes;
* ongoing or past medical treatments affecting wound healing, terminated less than 3 months prior to the study-related intervention

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Relative ratio between the detectable area covered by cement remnants per crown site and the total crown | Crowns were retrieved for analysis immediately after intraoral cementation and residual cement removal.
  Digital photographs of the specimens were obtained using custom-made equipment with a standardized distance. The images were analyzed as follows: the contours of the area covered by residual cement were identified visually after optical magnification and marked; the contours comprising the entire surface area of the prosthetic superstructure, i.e. abutment and crown, were determined; the ratio between the area covered with cement and the total surface area per aspect of the specimen was calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Eglė Vindašiūtė-Narbutė, Principal Investigator — Vilnius Implantology Center
Locations (1):
- Vilnius Implantology Center, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No